CLINICAL TRIAL: NCT05794633
Title: Effectiveness of Acupuncture Therapy in Patients With Subacromial Impingement Syndrome, Randomized Placebo-controlled Trial
Brief Title: Acupuncture Therapy in Patients With Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Karamanlıoğlu, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK-2012-70
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acupuncture; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients will be evaluated by the same physiatrist who are blinded to the randomization process and treatment protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental): The patients will be recieved two days a week for 8 sessions with sterile 25*40 mm needles.Selected points are as local points, 2 painful points (ahshi point) in the shoulder region, Large intestine 4, 15, Gallbladder 21, Triple warmer 5, 14 Small intestine 9; as distant points Gallbladder 34 and Stomach 38.
  Patients will recieve also exercise treatment for 8 weeks and coldpack for 4 weeks
  Interventions: Other: Acupuncture
- Placebo Acupuncture Group (Placebo Comparator): The patients will be recieved two days a week for 8 sessions with placebo needle. Selected points are Large intestine 15 Triple warmer 14 gallbladder 21 and small intestine 9. We will use the Placebo needle (blunt needle, tip obtuse, when acupuncture the feeling is similar to acupuncture needles into the skin, but it retracts instead of piercing the skin) to conduct acupuncture treatment. The retention time will be the same as those in the acupuncture group. The specialist will give the subjects verbal cues before and during the acupuncture manipulation, which further reduces the subjects' doubts about the authenticity of acupuncture in the this group. To ensure the implementation of the blinding method, all patients will be treated independently and avoid contacting with each other.
  Patients will recieve also exercise treatment for 8 weeks and coldpack for 4 weeks
  Interventions: Other: Placebo acupuncture

INTERVENTIONS:
Other: Acupuncture — The patients will be recieved two days a week for 8 sessions with sterile 25*40 mm needles.Selected points are as local points, 2 painful points (ahshi point) in the shoulder region, Large intestine 4, 15, Gallbladder 21, Triple warmer 5, 14 Small intestine 9; as distant points Gallbladder 34 and Stomach 38.
  Patients will recieve also exercise treatment for 8 weeks and coldpack for 4 weeks
  Arms: Acupuncture Group
Other: Placebo acupuncture — The patients will be recieved two days a week for 8 sessions with placebo needle. Selected points are Large intestine 15 Triple warmer 14 gallbladder 21 and small intestine 9. We will use the placebo needle (blunt needle, tip obtuse, when acupuncture the feeling is similar to acupuncture needles into the skin, but it retracts instead of piercing the skin) to conduct acupuncture treatment. The retention time will be the same as those in the acupuncture group. The specialist will give the subjects verbal cues before and during the acupuncture manipulation, which further reduces the subjects' doubts about the authenticity of acupuncture in the this group. To ensure the implementation of the blinding method, all patients will be treated independently and avoid contacting with each other.
  Patients will recieve also exercise treatment for 8 weeks and coldpack for 4 weeks
  Arms: Placebo Acupuncture Group

SUMMARY:
Shoulder pain is highly prevalent within general population, and shoulder impingement syndrome (SIS) is a common cause of shoulder pain. A small number of clinical and methodologically diverse trials have been published recently which show little evidence to support or refute the use of acupuncture for shoulder pain. Some researchers concluded, there is a need for further well-designed clinical trials. Our aim in this study is to investigate the effect of acupuncture treatment on pain, range of motion, functionality and quality of life in patients diagnosed with Subacromial Impingement Syndrome as a result of clinical and radiological tests.

DETAILED DESCRIPTION:
A randomized, prospective, double-blinded, placebo-controlled trial will be conducted. Patients diagnosed with shoulder impingement syndrome will be divided into two groups (acupuncture and placebo acupuncture) The evaluation will be performed at treatment initiation and at the end of the treatment and 1 month after treatment initiation.All patients will be evaluated by the same physiatrist who are blinded to the randomization process and treatment protocols.Primary outcome is pain which will be evaulated with visual analogue scale (VAS) for rest, activity, and sleep-disturbing. Secondary outcomes are shoulder range of motion in all groups will be evaluated with goniometer, shoulder function which will be evaulated with the Shoulder Pain and Disability Index (SPADI) and The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) and quality of life in all groups will be evaluated with The Western Ontario Rotator Cuff Index (WORC).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Subacromial impingement syndrome
* Age range from 20-65 years
* Pain VAS ≥ 4
* Shoulder impingement symptoms lasting at least 6 weeks

Exclusion Criteria:

* Presence of other shoulder pathologies
* Previous applications of physiotherapy and injection of hyaluronic acid and/or corticosteroid during the preceding 3 months;
* Presence of cervical pain or other conditions such as fibromyalgia confusing the clinical picture
* Presence of malignancy, blood disorder, neurologic, motor, and/or sensory deficit in the upper extremity;
* Pregnancy,
* Local anesthetic allergy
* Previous acupuncture treatment
* History of deformities, fractures, or surgery of the shoulder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 months
  All groups will be evaluated for shoulder pain with visual analogue scale (VAS) for rest, activity, and sleep-disturbing.
Shoulder Pain and Disability Index | 2 months
  All groups will be evaluated for shoulder function with the Shoulder Pain and Disability Index (SPADI). SPADI:The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. To answer the questions, patients place a mark on a 10cm visual analogue scale for each question. Higher results indicate worse function.
The Disabilities of the Arm, Shoulder and Hand Score | 2 months
  All groups will be evaluated for shoulder function with The Disabilities of the Arm, Shoulder and Hand Score (QuickDash). The QuickDASH only contains 11 items. It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level. Higher results indicate worse function.

SECONDARY OUTCOMES:
Shoulder range of motion | 2 months
  All groups will be evaluated for shoulder range of motion with goniometer.
Quality of life index | 2 months
  Quality of life: All groups will be evaluated for quality of life with The Western Ontario Rotator Cuff Index (WORC). Each item in WORC has a possible score from 0-100 (100mm VAS). Scores can be computed for individual subscales and summated for a total score, which can range from 0-2100, with a higher score representing lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Silte Karamanlioglu, Principal Investigator — Fatih Sultan Mehmet Traning and Research Hospital; Meryem Yilmaz Kaysin, Study Chair — Fatih Sultan Mehmet Traning and Research Hospital; Feyza Akan Begoglu, Study Chair — Fatih Sultan Mehmet Traning and Research Hospital; Pinar Akpinar, Study Chair — Fatih Sultan Mehmet Traning and Research Hospital; Feyza Unlu Ozkan, Study Chair — Fatih Sultan Mehmet Traning and Research Hospital; Ilknur Aktas, Study Chair — Fatih Sultan Mehmet Traning and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karamanlioglu DS, Kaysin MY, Begoglu FA, Akpinar P, Ozkan FU, Aktas I. Effects of acupuncture on pain and function in patients with subacromial impingement syndrome: A randomized sham-controlled trial. Integr Med Res. 2024 Jun;13(2):101049. doi: 10.1016/j.imr.2024.101049. Epub 2024 May 25. PMID 38948487